CLINICAL TRIAL: NCT04422041
Title: Comparison of Early Versus Very Early Postnatal Discharge on Hospital Readmissions in Newborns: A Prospective Study
Brief Title: Comparison of Early Versus Very Early Postnatal Discharge on Hospital Readmissions in Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, Erika Ochoa-Correa, Professor, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PE15-039
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Hospital Readmission; Newborn Morbidity; Newborn Complication; Newborn
Keywords: Newborn Infant; Hospital readmission; Early discharge; Very early discharge

STUDY DESIGN:
Intervention Model Description: They were selected based on a random computer program in a 1: 1 model, assigning each subject randomly to one of the two study groups
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors consisted of hospital staff not involved in the investigation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early discharge (Active Comparator): Discharge between 24 and 48 hours
  Interventions: Other: Discharge time between 24 and 48 hours
- Very early discharge (Experimental): Discharge in less than 24 hours
  Interventions: Other: Time to discharge less than 24 hours

INTERVENTIONS:
Other: Time to discharge less than 24 hours — Allow the joint medical discharge of the newborn together with its mother in less than 24 hours after birth in a healthy patient, without obstetric complications and who does not present comorbidities and complications.
  Arms: Very early discharge
Other: Discharge time between 24 and 48 hours — Allow the joint medical discharge of the newborn together with its mother between 24-48 hours after birth in a healthy patient, without obstetric complications and who does not present comorbidities and complications.
  Arms: Early discharge

SUMMARY:
This study compared hospital readmission and complications between very early discharge and early discharge in healthy newborn patients.

DETAILED DESCRIPTION:
Introduction. Very early postnatal discharge is defined as a hospital stay of the mother-child dyad of less than 24 hours. It is usually performed in public institutions of low-income countries due to high birth rates; it has not been associated to a higher proportion of neonatal admissions, however, very early discharge might increase this risk. The objective of this study was to compare the rate hospital readmission in patients with very early vs early postnatal discharge.

Methods A prospective, randomized clinical study was performed with healthy term infants born in a hospital in Mexico from July 2016 to June 2018. Sample was randomized into two groups, a very early discharge group (<24 hours) and an early discharge group (24-48 hours). Hospital readmission rate was analyzed in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy newborns that were born from vaginal delivery in primiparous or multiparous women where both the mother and the newborn were deemed as eligible for early discharge according to the American Association of Pediatrics criteria and by a clinical obstetric mother evaluation.

Exclusion Criteria:

* Placenta praevia, abnormal bleeding during vaginal delivery (considered as greater than 500mL), inhability to deambulate, medical complications from previous a previous pregnancy, 3rd or 4th degree perineal laceration as well as medical conditions that required any monitorization for more than 24 hours after delivery.

Ages: 1 Minute to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 354 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-07-29 (Actual)

PRIMARY OUTCOMES:
Hospital readmission rate | 28 days
  Proportion of participant newborns who were readmitted into the hospital during follow up

SECONDARY OUTCOMES:
Rate of attention in emergency services | 28 days
  Proportion of participant newborns who attended the emergency services during follow up
Readmission rate associated factors | 28 days
  Statistical associations between the primary outcome and other variables of interest

CONTACTS AND LOCATIONS:
Overall Officials: Erika Ochoa-Correa, M.D., Principal Investigator — Universidad Autonoma de Nuevo Leon, School of Medicine, Department of Pediatrics

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones E, Taylor B, MacArthur C, Pritchett R, Cummins C. The effect of early postnatal discharge from hospital for women and infants: a systematic review protocol. Syst Rev. 2016 Feb 8;5:24. doi: 10.1186/s13643-016-0193-9. PMID 26857705
- [Background] Brown S, Small R, Faber B, Krastev A, Davis P. Early postnatal discharge from hospital for healthy mothers and term infants. Cochrane Database Syst Rev. 2002;(3):CD002958. doi: 10.1002/14651858.CD002958. PMID 12137666
- [Background] Benitz WE; Committee on Fetus and Newborn, American Academy of Pediatrics. Hospital stay for healthy term newborn infants. Pediatrics. 2015 May;135(5):948-53. doi: 10.1542/peds.2015-0699. PMID 25917993
- [Background] Chalmers B, Mangiaterra V, Porter R. WHO principles of perinatal care: the essential antenatal, perinatal, and postpartum care course. Birth. 2001 Sep;28(3):202-7. doi: 10.1046/j.1523-536x.2001.00202.x. PMID 11552969
- [Background] Capurro H, Konichezky S, Fonseca D, Caldeyro-Barcia R. A simplified method for diagnosis of gestational age in the newborn infant. J Pediatr. 1978 Jul;93(1):120-2. doi: 10.1016/s0022-3476(78)80621-0. No abstract available. PMID 650322
- [Background] SILVERMAN WA, ANDERSEN DH. A controlled clinical trial of effects of water mist on obstructive respiratory signs, death rate and necropsy findings among premature infants. Pediatrics. 1956 Jan;17(1):1-10. No abstract available. PMID 13353856
- See also: Norma Oficial Mexicana NOM-007-SSA2-2016 para la atención de la mujer durante el embarazo, parto y puerperio, y de la persona recién nacida. — http://www.cndh.org.mx/sites/all/doc/Programas/VIH/Leyes%20y%20normas%20y%20reglamentos/Norma%20Oficial%20Mexicana/NOM-007-SSA2-2016%20Embarazo,%20parto%20y%20puerperio.pdf